CLINICAL TRIAL: NCT04665778
Title: Prediction of the Patient Pathway in Emergency Room in an Exceptional Sanitary Situation
Acronym: 3PU-SSE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0055
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Emergencies
Keywords: Covid19; patient flow; emergency overcrowding
MeSH Terms: conditions — COVID-19; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high risk of hospitalization
  Interventions: Other: hospital bedroom booking
- not high risk of hospitalization

INTERVENTIONS:
Other: hospital bedroom booking — Patient in high risk of hospitalization group benefits a dedicated process to find and book a bedroom
  Groups: high risk of hospitalization

SUMMARY:
The COVID-19 outbreak leads to optimize the pathway in emergency departments. The length of time spent in the Emergency Department is linked to the morbi-mortality and the risk of COVID-19 transmission. The Amiens-Picardy University Hospital has developed an application (3P-U) that optimizes patient flow. It identifies the need of hospitalization and problems on the care path. Patients are categorized in high risk or not high probabilty of hospitalization. The main goal of this project is to evaluate the impact on the patient flow of the 3P-U application. Early lookup of bed for high probability hospitalization should be linked to a reduced time of length. This study will compare the time of length between this both groups.

ELIGIBILITY:
Inclusion Criteria:

* every patient that consults in the Adult Emergency Department

Exclusion Criteria:

* patients directly transferred to Intensive Care Units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that consults in adult emergency department should be included
Sampling Method: Non-Probability Sample
Enrollment: 1516 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Variation of the length of stay between high probability of hospitalization group and not high risk of hospitalization group. | up to 3 months
  Variation of the length of stay between high probability of hospitalization group and not high risk of hospitalization group.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No